CLINICAL TRIAL: NCT04591249
Title: Developing a Novel Physical Activity Intervention for Patients Following Lumbar Spine Surgery (PASS Trial)
Brief Title: Physical Activity Intervention for Patients Following Lumbar Spine Surgery
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Hiral Master, Post-doctoral Research Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201126
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Spinal Degenerative Disorder; Spinal Stenosis; Spondylosis
Keywords: physical activity; wearable technology; behavioral model; funciton; disability; pain
MeSH Terms: conditions — Spinal Stenosis; Spondylosis; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Two-group, single-center randomized, controlled study in 30 patients undergoing spine surgery for a lumbar degenerative condition to examine the feasibility and acceptability of an 8-week remote physical activity intervention.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual postoperative care (Other): Participants randomized to usual care group will receive postoperative care as determined by their treating surgeon.
  Interventions: Other: Usual care
- Usual postoperative care + Physical activity intervention (Experimental): Participants randomized to the physical activity intervention group will receive usual postoperative care as determined by their treating surgeon and novel physical activity intervention.
  Interventions: Behavioral: Physical activity intervention; Other: Usual care

INTERVENTIONS:
Behavioral: Physical activity intervention — Participants will 1) receive Fitbit, 2) be enrolled in a secure electronic platform to access Fitbit data, 3) receive 8-week remote counseling by a physical therapist that will include motivational interviewing and creating SMART goals (1 session per week) through a web-based teleconference platform, and 4) receive usual postoperative care directed by their surgeon. The first session will be 45 minutes and sessions 2-8 will be 30 minutes each. During the sessions, participant's confidence in meeting daily step goals will be assessed using a 0-10 scale. If self-reported confidence to meet their goal is <8, the physical therapist will help participants modify their goal using techniques such as problem-solving, positive statements and affirmations. Progression will be made only if daily steps goals are met for at least 4 out of 7 days a week. If this weekly step goal is not met, a physical therapist will help the participant identify solutions for realistic progression.
  Arms: Usual postoperative care + Physical activity intervention
Other: Usual care — Participants will receive postoperative care as determined by their treating surgeon. This includes lifting restrictions, advice to stay active, and oral analgesics as needed. Physical therapy referral will be at the discretion of the surgeon. However, physical therapy is not typically started until 12 weeks after surgery.

SUMMARY:
There is a critical need to target physical activity during postoperative management to optimize long-term recovery after lumbar spine surgery. The overall objective of this study is to conduct a two-group randomized control trial (RCT) to examine the feasibility and acceptability of a physical activity telehealth intervention delivered by a physical therapist for improving disability, physical function, pain, and physical activity compared to usual care after spine surgery for a degenerative lumbar condition. The physical activity intervention will include wearable technology and remote physical therapist support to counsel patients on a realistic progression of physical activity (steps per day). The central hypothesis is that this 8-week physical activity intervention performed at two weeks after surgery will be feasible and acceptable. The results of our randomized trial will be used to support a large multi-site clinical trial to test the effectiveness and implementation of this intervention

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 years or older, of both sexes and all races
2. Scheduled for surgical treatment of a lumbar degenerative condition (spinal stenosis, spondylosis with or without myelopathy, and degenerative spondylolisthesis) using laminectomy with or without arthrodesis (i.e., fusion) procedures.
3. Participants will be English speaking due to the feasibility of employing study personnel to deliver and assess the study intervention.

Exclusion Criteria:

1. Patients having microsurgical techniques as the primary procedure, such as an isolated laminotomy or microdiscectomy will be excluded because individuals having these minimally invasive surgical techniques tend to have a less severe case of lumbar degeneration.
2. Patients having surgery for spinal deformity as the primary indication or surgery secondary to pseudarthrosis, trauma, infection, or tumor
3. Prior history of lumbar spine surgery
4. Presence of back and/or lower extremity pain < 3 month
5. History of neurological disorder, resulting in moderate to severe movement dysfunction
6. Unable to provide stable address and access to a telephone indicating the inability to participate in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | At 2 weeks after spine surgery
  Proportion of potential eligible participants successfully contacted who agreed to participate and randomized.
Adherence rate to study protocol at 3 months after spine surgery | From 2 weeks to 3-months after spine surgery
  Proportion of participants who will complete the assessment at 2 weeks and 3 months after spine surgery.
Adherence rate to study protocol at 6 months after spine surgery | From 2 weeks to 6-months after spine surgery
  Proportion of participants who will complete the assessment at 2 weeks and 6 months after spine surgery.
Adherence to physical activity intervention | From 2-weeks to 3-months after spine surgery
  Number of weekly step goals completed by participant, which will be examined via Fitabase.
  In addition, number of weekly Zoom calls completed with the physical therapist will be recorded
Number of adverse events | From 2-weeks to 3-months after spine surgery
  During the intervention phase, the study physical therapist will document adverse events related to walking to assess safety.

SECONDARY OUTCOMES:
Oswestry Disability Index | Preoperative, and at 2 weeks (baseline), 3-, and 6-months after spine surgery
  A 10-item questionnaire will be used to measure condition-specific disability that assesses the impact of lumbar spinal disorders on activities of daily living. Each item is measured from 0 to 5, representing low and high disability, respectively. Total score ranges from 0 to 50.
PROMIS Physical Function | Preoperative, and at 2 weeks (baseline), 3-, and 6-months after spine surgery
  PROMIS Physical Function 4-item short form will be used to measure physical function. Each item is measured from 1 to 5, representing low to high physical function, respectively. Total score ranges from 4 to 20.
Numeric rating scale for back pain | Preoperative, and at 2 weeks (baseline), 3-, and 6-months after spine surgery
  Numeric rating scale will be used to assess the pain intensity using the single-item for back, which is scored from 0 to 10, representing no pain and the worst pain, respectively.
Numeric rating scale for leg pain | Preoperative, and at 2 weeks (baseline), 3-, and 6-months after spine surgery
  Numeric rating scale will be used to assess the pain intensity using the single-item for leg, which is scored from 0 to 10, representing no pain and the worst pain, respectively.
Intensity of physical activity | Preoperative, and at 2 weeks (baseline), 3-, and 6-months after spine surgery
  A research-grade triaxial accelerometer (Actigraph GT3x) will be used to quantify time spent in different intensities of physical activity per day.
Physical activity volume | Preoperative, and at 2 weeks (baseline), 3-, and 6-months after spine surgery
  A research-grade triaxial accelerometer (Actigraph GT3x) will be used to quantify total number of steps per day.
Depressive symptoms | Preoperative, and at 2 weeks (baseline), 3-, and 6-months after spine surgery
  PROMIS Depression 4 item short form will be used to measure depressive symtpoms. Each item is measured from 1 to 5, representing low to high depressive symptoms. Total score ranges from 4 to 20.
Fear of movement | Preoperative, and at 2 weeks (baseline), 3-, and 6-months after spine surgery
  A 13-item Tampa Scale for Kinesiophobia will be used to measure fear of movement. It has two sub-scales (activity avoidance and fear of pain) and the total score ranges from 13 to 52 with higher scores indicating greater fear of movement.

OTHER OUTCOMES:
Opioid Use | Preoperative, and at 2 weeks (baseline), 3-, and 6-months after spine surgery
  A single-item Patient-reported opioid use questionnaire (yes vs. no).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin R Archer, DPT, PhD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Given the pilot nature of the trial, the IPD will not be available to other researchers.

REFERENCES:
- See also: Website that provides brief description of the PASS trial — https://www.vumc.org/musculoskeletal-research/spine